CLINICAL TRIAL: NCT06462443
Title: A Prospective Study of RISE (Resilience, Insight, Self-compassion, Empowerment) for Physicians
Brief Title: A Prospective Study of RISE for Physicians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2057666
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-07

CONDITIONS: Stress; Burn Out
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: Single group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Intervention group will attend the RISE for Physicians program, a 2.5 day retreat-style psychoeducational group program facilitated by licensed mental health professionals (LMHPs)
  Interventions: Behavioral: RISE for Physicians Program

INTERVENTIONS:
Behavioral: RISE for Physicians Program — RISE for Physicians Program. Psychoeducational group program designed to impact resilience, insight, self-compassion, and empowerment

SUMMARY:
The purpose of this study is to determine whether the RISE for Physicians program has a significant impact on physicians' burnout, resilience, insight, self-compassion, empowerment, and professional and personal mental health and well-being.

DETAILED DESCRIPTION:
This study will include 36 subjects recruited from employed physicians and non-employed physicians with privileges at AdventHealth. The study will include data collection along with program participation. Program will consist of a 2.5 day retreat facilitated by a licensed mental health professional. Data collection will be at 3 timepoints and include 10 surveys that are expected to take 30 minutes to complete.

ELIGIBILITY:
Inclusion Criteria:

* AdventHealth employed or contract physician
* Or non-employed physician with AdventHealth privileges (hospital, emergency room, or AHMG practice)

Exclusion Criteria:

* A resident physician
* Advanced practice provider
* Executive leader

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2025-11-12 (Actual); Study Completion 2025-11-12 (Actual)

PRIMARY OUTCOMES:
Maslach Burnout Inventory - Human Services Survey | Baseline, 1-month follow-up, 3-month follow-up
  22-item questionnaire with the following response categories: 0=never, 1=a few times a year or less, 2=once a month or less, 3=a few times a month, 4=once a week, 5=a few times a week, 6=every day

SECONDARY OUTCOMES:
Professional Quality of Life Scale | Baseline, 1- and 3-month follow-up
  30-item questionnaire with the following response categories: 1=never, 2=rarely, 3=sometimes, 4=often, 5=very often
Brief Resilience Scale | Baseline, 1- and 3-month follow-up
  6-item questionnaire with the following response categories: 1=strongly agree, 2=disagree, 3=neutral, 4=agree, 5=strongly agree
Self-Reflection and Insight Scale - Short Form | Baseline, 1- and 3-month follow-up
  12-item questionnaire with the following response categories: 1=strongly disagree, 2, 3, 4, 5, 6, 7=strongly agree
Self-Compassion Scale - Short Form | Baseline, 1- and 3-month follow-up
  12-item questionnaire with the following response categories: 1=almost never, 2, 3, 4, 5=almost always
General Self-Efficacy Scale | Baseline, 1- and 3-month follow-up
  10-item questionnaire with the following response categories: 1=not at all true, 2=barely true, 3=moderately true, 4=exactly true
Perceived Stress Scale | Baseline, 1- and 3-month follow-up
  10-item questionnaire with the following response categories: 0=never, 1=almost never, 2=sometimes, 3=fairly often, 4=very often
Work-Life Climate Scale | Baseline, 1- and 3-month follow-up
  7-item questionnaire with the following response categories: rarely or none of the time (<1 day), some or a little of the time (1-2 days), occasionally or a moderate amount of time (3-4 days), all of the time (5-7 days)
Moral Injury Outcomes Scale | Baseline, 1- and 3-month follow-up
  14-item questionnaire with the following response categories: 0=strongly agree, 1=disagree, 2=neither agree or disagree, 3=agree, 4=strongly agree
Generalized Anxiety Disorder - 2 item scale | Baseline, 1- and 3-month follow-up
  2-item questionnaire with the following response categories: 0=not at all, 1=several days, 2=more than half the days, 3=nearly every day
Patient Health Questionnaire - 2 item | Baseline, 1- and 3-month follow-up
  2-item survey with the following response categories: 0=not at all, 1=several days, 2=more than half the days, 3=nearly every day

CONTACTS AND LOCATIONS:
Overall Officials: Amanda T Sawyer, PhD, Principal Investigator — AdventHealth
Locations (1):
- AdventHealth, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bailey AK, Sawyer AT, Robinson PS. A Psychoeducational Group Intervention for Nurses: Rationale, Theoretical Framework, and Development. J Am Psychiatr Nurses Assoc. 2023 May-Jun;29(3):232-240. doi: 10.1177/10783903211001116. Epub 2021 Jun 22. PMID 34154451
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Kroenke K, Spitzer RL, Williams JB, Monahan PO, Lowe B. Anxiety disorders in primary care: prevalence, impairment, comorbidity, and detection. Ann Intern Med. 2007 Mar 6;146(5):317-25. doi: 10.7326/0003-4819-146-5-200703060-00004. PMID 17339617
- [Background] Kroenke K, Spitzer RL, Williams JB. The Patient Health Questionnaire-2: validity of a two-item depression screener. Med Care. 2003 Nov;41(11):1284-92. doi: 10.1097/01.MLR.0000093487.78664.3C. PMID 14583691
- [Background] Litz BT, Plouffe RA, Nazarov A, Murphy D, Phelps A, Coady A, Houle SA, Dell L, Frankfurt S, Zerach G, Levi-Belz Y; Moral Injury Outcome Scale Consortium. Defining and Assessing the Syndrome of Moral Injury: Initial Findings of the Moral Injury Outcome Scale Consortium. Front Psychiatry. 2022 Jul 5;13:923928. doi: 10.3389/fpsyt.2022.923928. eCollection 2022. PMID 35873252
- [Background] 6. Maslach C, Jackson SE, Leiter MP. Maslach Burnout Inventory manual, 3rd ed. Palo Alto, CA: Consulting Psychologists Press, 1996.
- [Background] Raes F, Pommier E, Neff KD, Van Gucht D. Construction and factorial validation of a short form of the Self-Compassion Scale. Clin Psychol Psychother. 2011 May-Jun;18(3):250-5. doi: 10.1002/cpp.702. Epub 2010 Jun 8. PMID 21584907
- [Background] Sawyer AT, Bailey AK, Green JF, Sun J, Robinson PS. Resilience, Insight, Self-Compassion, and Empowerment (RISE): A Randomized Controlled Trial of a Psychoeducational Group Program for Nurses. J Am Psychiatr Nurses Assoc. 2023 Jul-Aug;29(4):314-327. doi: 10.1177/10783903211033338. Epub 2021 Jul 23. PMID 34293934
- [Background] Sawyer AT, Tao H, Bailey AK. The Impact of a Psychoeducational Group Program on the Mental Well-Being of Unit-Based Nurse Leaders: A Randomized Controlled Trial. Int J Environ Res Public Health. 2023 Jun 2;20(11):6035. doi: 10.3390/ijerph20116035. PMID 37297639
- [Background] 10. Schwarzer, R., & Jerusalem, M. (1995). Generalized Self-Efficacy Scale. J. Weinman, S. Wright, & M. Johnston, Measures in health psychology: A user's portfolio. Causal and control beliefs, 35, 37.
- [Background] 11. Silva PJ. The Self-Reflection and Insight Scale: Applying item response theory to craft an efficient short form. Curr Psychol. 2022;41:8635-8645. doi:10.1007/s12144-020-01299-7
- [Background] Smith BW, Dalen J, Wiggins K, Tooley E, Christopher P, Bernard J. The brief resilience scale: assessing the ability to bounce back. Int J Behav Med. 2008;15(3):194-200. doi: 10.1080/10705500802222972. PMID 18696313
- [Background] 13. Stamm, B. H. (2010). Professional Quality of Life: Compassion Satisfaction and Fatigue Version 5 (ProQOL). http://www.proqol.org.